CLINICAL TRIAL: NCT03806998
Title: Effects of a Ketoacid Supplementation on Urinary Urea Nitrogen Excretion in Patients With Stage III to IV Renal Failure
Brief Title: Effects of a Ketoacid Supplementation in Patients With Stage III to IV Renal Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Servicio de Salud Metropolitano Oriente (Unknown)
Responsible Party: Principal Investigator, Eduardo Lorca, Chief Cardiovascular Program, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ketosterilrenal
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Keto Acids

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assgned to receive the ketoacid supplement or placebo
Who Masked: Participant
Masking Description: There will be no masking of the treatment arm for researchers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketoacid supplementation (Experimental): Will receive a ketoacid supplement containing 630 mg of ketoacids in a dose of 1 tablet every 5 kg of body weight
  Interventions: Dietary Supplement: Ketoacids
- Placebo (Placebo Comparator): Will receive placebo tablets in a dose of 1 tablet every 5 kg of body weight
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketoacids — Provision of 1 Tablet containing 630 mg of ketoacids every 5 kg of body weight during 16 weeks
  Arms: Ketoacid supplementation
Dietary Supplement: Placebo — Provision of placebo capsules similar to active supplement
  Arms: Placebo

SUMMARY:
The aim of the study is to demonstrate that a ketoacid supplement in patients with stage III to IV chronic renal failure, reduces the excretion of urinary urea nitrogen

DETAILED DESCRIPTION:
Patients with an estimated glomerular filtration rate of less than 25 ml/kg/min, not on renal substitution therapy, without important concomitant diseases and aged between 40 and 70 years, will be invited to participate in the study. They will be randomly assigned to a group that will receive receive a supplement of ketoacids (Ketosteril) 1 tablet containing 630 mg of ketoacids every 5 kg of body weight and a diet containing 25 to 35 kcal/kg and 0.3 g/protein per day or to a group receiving placebo and a diet containing 25 to 35 kcal/kg and 0.6 g/protein per day. The intervention will last 16 weeks. At baseline and the end of the intervention a blood sample will be obtained to measure creatinine, urea nitrogen and cystatin C. Also a spot urine sample will be obtained to measure urea nitrogen and creatinine excretion. The compliance with the dietary prescription and the ketoacid or placebo supplement will be assessed every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate of less tan 25/ml/min/1.73m2
* Not on renal substitution therapy
* Absence of severe life threatening concomitant diseases

Exclusion Criteria:

* Malignant or renovascular hypertension
* Use of systemic steroids or immunosuppressant drugs
* Alcohol or illicit drug abuse
* A body mass index of less tan 18 kg/m2

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate | 16 weeks
  glomerular filtration rate estimated using the CKD-EPI formula for Cystatin-C
Urinary urea nitrogen excretion | 16 weeks
  Measurement of urea nitrogen i na spot urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bunout, MD, Principal Investigator — INTA University of Chile
Locations (1):
- Hospital del Salvador, Santiago, Santiago Metropolitan, Chile